CLINICAL TRIAL: NCT06403852
Title: Investigating Near-Threshold Perception During Anesthetic Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zirui Huang, Research Assistant Professor, Anesthesiology and Research Fellow, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00251768; R01GM103894 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Propofol; Anesthesia; fMRI
Keywords: Hypnotics and Sedatives; Central Nervous System Depressants; Physiological Effects of Drugs; Anesthetics, Intravenous; Anesthetics, General; Anesthetics; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Image recognition task (Experimental): The stimulus set will include real and scrambled images, where the scrambled images will be created by phase-shuffling a randomly chosen real image from each category to preserve category specific low-level image features. Each object category will include four unique real images and one scrambled image. Each image will be repeated 10 times (i.e., trials) for each 16-min session. The pre-stimulus interval will vary randomly from trial to trial between 4 and 8 seconds to prevent stimulus timing predictability. The stimuli will be presented in a randomized order to prevent category predictability.
  Interventions: Combination Product: Functional Magnetic Resonance Imaging (fMRI) with propofol

INTERVENTIONS:
Combination Product: Functional Magnetic Resonance Imaging (fMRI) with propofol — Three 16-min sessions in wakeful baseline, light sedation, and recovery will be conducted (Fig. 2). Light sedation will be achieved by IV infusion of propofol to achieve effect-site concentrations of 1.0 μg/ml. Infusion rate will be manually controlled. An initial bolus dose (525 µg/kg) and subsequent infusion rate (82 µg/kg/min) for each participant

SUMMARY:
The researchers expect to gain a deeper understanding of mental function during different levels of anesthesia, and to evaluate if the use of ultrasonic brain stimulation accelerates return to consciousness.

Propofol is FDA approved for use in patients undergoing an anesthetic for medical treatment but is not approved for use in healthy volunteers.

DETAILED DESCRIPTION:
The stimulus set will include real and scrambled images, where the scrambled images will be created by phase-shuffling a randomly chosen real image from each category to preserve category specific low-level image features. Because scrambled images do not include an object stimulus, the images are used as "catch trials" to determine the subjects' baseline tendency to give positive responses to a question about the subjects' recognition experience. Each object category will include four unique real images and one scrambled image. Each image will be repeated 10 times (i.e., trials) for each 16-min session. The pre-stimulus interval will vary randomly from trial to trial between 4 and 8 seconds to prevent stimulus timing predictability. The stimuli will be presented in a randomized order to prevent category predictability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy study subjects with American Society of Anesthesiologists (ASA)-1 status.
* Right-handed
* Body mass index (BMI) less than 30.
* All subjects will be English speakers.

Exclusion Criteria:

* Medical contraindication to magnetic resonance imaging (MRI) scanning; are unable to undergo MRI scanning because of possible pregnancy or currently breastfeeding, BMI>30, metallic substances in the body, claustrophobia, anxiety, or cardiopulmonary disease; or have an intracranial structural abnormality on T1-weighted MRI scans.
* History of allergy to propofol, eggs or egg products, soybean or soybean products, neurological, cardiovascular, or pulmonary illness; significant head injury with loss of consciousness; learning disability or other developmental disorder; sleep apnea or any severe snoring history; gastroesophageal reflux disease (GERD) or heartburn; pancreatitis or a history of pancreatitis, or sensory/motor loss sufficient to interfere with performance of the study.
* Tattoos in the head or neck region will be excluded from study; other tattoos are subject to determination by investigators based on their assessment regarding participant safety. To eliminate aspiration risk subjects will also be excluded if they have had recent food or liquid intake (within 8 hours).
* History of drug use, have a positive drug screen, are unwilling to abstain from alcohol for 24 hours prior to dosing, or have a current history of nicotine use.
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) response to visual stimuli | Up to 90 minutes
  Visual stimuli evoked activity was quantified by measurements of the fMRI BOLD signal. Neural response to a natural visual stimulus will be assessed during both conscious and anesthetized states.

SECONDARY OUTCOMES:
Perceptual criterion (c) derived from the Signal Detection Theory (SDT) | Up to 90 minutes
Sensitivity (d') criterion derived from the Signal Detection Theory (SDT) | Up to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zirui Huang, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT06403852/ICF_001.pdf